CLINICAL TRIAL: NCT01264614
Title: Neuropsychological and Neuroimaging Effects of Strengthening Exercise for Early Dementia and Normative Older Adults
Brief Title: Effects of Strengthening Exercise on the Brain for Early Dementia and Normative Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Union College, New York (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Cay Anderson-Hanley, Principal Investigator, Union College, New York
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIRB#00663
Record Dates: First submitted 2010-12-21; First posted 2010-12-22 (Estimated); Results first posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Cognitive Decline; Dementia; Alzheimer's Disease; Mild Cognitive Impairment
Keywords: exercise; neuropsychological; dementia; Alzheimer's Disease; mild cognitive impairment; strength; MCI; AD; EEG; neurophysiological; growth factor; cognitive decline; executive function
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Alzheimer Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early stage dementia (Experimental): Individuals with early stage dementia who attended a Adult Day Care Program at least twice a week. Participants engaged in a strengthening exercise program three to five times per week for 10 weeks.
  Interventions: Behavioral: Strengthening exercise
- Normative older adults (Active Comparator): Normative older adults with no known neurological condition. Participants engaged in a strengthening exercise program three to five times per week for 10 weeks.
  Interventions: Behavioral: Strengthening exercise

INTERVENTIONS:
Behavioral: Strengthening exercise — 3 months of 3-5 times per week of low-intensity exercises using a chair and small weights
  Other Names: Strong Bones Program

SUMMARY:
This study will evaluate the effects of low-intensity strengthening exercise on the brain (thinking and processing speed) for patients with early dementia, compared with normative older adults. Participants will engage in 3 months of exercise 3-5 times per week using a chair and small weights. It is hypothesized that there will be a significant improvement in brain function.

DETAILED DESCRIPTION:
1. Objective(s): This study will evaluate the neuropsychological and neurophysiological effects of low-intensity strengthening exercise for patients with early dementia, compared with normative older adults.
2. Research Design: This is a quasi-experimental design in which change over time as a result of the exercise intervention will be compared with change over time seen in a normative sample.
3. Methodology: The aim is to enroll 12 participants with early dementia and 12 normative controls, all who are interested in starting a strengthening exercise program. Neuropsychological evaluation, resting electroencephalography (EEG), and event-related potentials (ERP) data collection will commence prior to the start of exercise. Participants will participate in an exercise class 2-3x/wk for three months. Repeat neuropsychological, EEG, and ERP evaluations will occur at the conclusion of three months of exercise. The exercises consist of low-intensity exercises, using a chair and small weights. A leader trained in the Tufts University exercise model will conduct the classes.
4. Findings: The investigators hypothesize a positive impact of exercise on neuropsychological function, especially performance on tasks requiring executive functions. This change will be compared with performance of normative controls who also exercise. Changes in brain function will be explored using EEG and ERP, and results are expected to be similar to prior research examining older adult exercisers which shows improvement in function.

ELIGIBILITY:
Inclusion Criteria:

* Adult Day Program Participants with early dementia able to consent or assent with surrogate permission
* Control participants (55-100+ yo) able to participate at location with doctor permission

Exclusion Criteria:

* history of significant TBI, psychiatric condition, substance abuse, physical conditions that preclude participation in cognitive testing or strengthening exercises

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cay Anderson-Hanley, PhD, Principal Investigator — Union College
Locations (1):
- Stratton VA Medical Center, Albany, New York, United States

REFERENCES:
- [Result] Yerokhin V, Anderson-Hanley C, Hogan MJ, Dunnam M, Huber D, Osborne S, Shulan M. Neuropsychological and neurophysiological effects of strengthening exercise for early dementia: a pilot study. Neuropsychol Dev Cogn B Aging Neuropsychol Cogn. 2012;19(3):380-401. doi: 10.1080/13825585.2011.628378. Epub 2011 Dec 2. PMID 22136405

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Early stage dementia participants were drawn from the Adult Day Care Program (ADCP) at a Veterans Affairs Medical Center (VAMC) in the northeast United States. Normative older adult participants were either employees or volunteers at the same facility recruited by fliers.
Groups:
- Early Stage Dementia: Individuals with early stage dementia who attended a Adult Day Care Program at least twice a week.
- Normative Older Adults: Normative older adults with no known history of neurological condition.
Period: Overall Study
Arm/Group | Early Stage Dementia | Normative Older Adults
Started | 13 | 9
Completed | 12 | 7
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Population: 13 early dementia participants and 9 normative older adult participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Stage Dementia | Normative Older Adults | Total
Number analyzed (Participants) | 13 | 9 | 22
Age, Continuous [Mean (Full Range); unit: years] | 79.3 [60 to 95] | 62.8 [55 to 78] | 71.5 [55 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 13 | 8 | 21
Region of Enrollment [Number; unit: participants]
  United States | 13 | 9 | 22
Education [Mean (Full Range); unit: years] | 11.5 [6 to 16] | 11.6 [8 to 13] | 11.6 [6 to 16]

OUTCOME MEASURES:

1. Primary Outcome: Stroop Test Performance From Pre- to Post-intervention
Description: Average raw cognitive scores before (T1) and after (T2) strengthening exercise intervention. Lower scores on Stroop C (possible range 0-240 sec) represents better performance).
Time Frame: Baseline and 3 months
Population: Two of 9 normative participants, had to be dropped from analyses due to limited participation in the exercise program (less than once per week on average; health problems and snowy weather were the main limiting factors) and one dementia exerciser was dropped because he did not complete any of the outcome measures.
Measure: Mean (Standard Deviation); unit: Time to complete (seconds)
Arm/Group | Early Stage Dementia | Normative Older Adults
Number analyzed (Participants) | 12 | 7
Time to complete (seconds)
  Stroop C pre | 137.67 (102.30) | 56.17 (10.34)
  Stroop C post | 116.51 (64.44) | 55.13 (11.08)

2. Primary Outcome: Digits Backwards Test Performance From Pre- to Post-intervention
Description: Average raw cognitive scores before (T1) and after (T2) strengthening exercise intervention. Higher scores represent better performance (Digits backwards possible score range is 0-14 points).
Time Frame: Baseline and 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Early Stage Dementia | Normative Older Adults
Number analyzed (Participants) | 12 | 7
Points
  Digits Backward pre | 4.10 (1.73) | 5.50 (2.59)
  Digits Backward post | 3.90 (1.10) | 6.83 (2.71)

3. Primary Outcome: Color Trails Test Performance From Pre- to Post-intervention
Description: Average raw cognitive scores before (T1) and after (T2) strengthening exercise intervention. Higher scores represent better performance (Color Trails possible score range is 0-300 seconds).
Time Frame: Baseline and 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Time to complete (seconds)
Arm/Group | Early Stage Dementia | Normative Older Adults
Number analyzed (Participants) | 12 | 7
Time to complete (seconds)
  Color Trails 2 pre | 250.00 (186.45) | 124.00 (67.97)
  Color Trails 2 post | 259.01 (197.63) | 96.11 (19.97)

4. Primary Outcome: Fuld Test Performance From Pre- to Post-intervention
Description: Average raw cognitive scores before (T1) and after (T2) strengthening exercise intervention. Higher scores represent better performance (Fuld Semantic Recall possible score range is 0-20 points; Fuld Immediate and Delayed Recall possible score range is 0-10).
Time Frame: Baseline and 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Early Stage Dementia | Normative Older Adults
Number analyzed (Participants) | 12 | 7
Points
  Fuld Semantic Recall pre | 10.60 (3.66) | 18.80 (8.76)
  Fuld Semantic Recall post | 10.60 (4.27) | 18.60 (5.86)
  Fuld Immediate Recall pre | 2.90 (2.38) | 6.60 (1.34)
  Fuld Immediate Recall post | 4.40 (1.65) | 7.60 (1.52)
  Fuld Delayed Recall pre | 2.60 (2.41) | 8.40 (1.14)
  Fuld Delayed Recall post | 4.50 (2.72) | 8.20 (.45)

5. Primary Outcome: Figure Copy & Delayed Test Performance From Pre- to Post-intervention
Description: Average raw cognitive scores before (T1) and after (T2) strengthening exercise intervention. Higher scores represent better performance (Figure Copy & Delayed possible score range is 0-36 points).
Time Frame: Baseline and 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Early Stage Dementia | Normative Older Adults
Number analyzed (Participants) | 12 | 7
Points
  Figure Copy pre | 16.44 (6.96) | 28.67 (3.99)
  Figure Copy post | 22.06 (9.96) | 30.33 (3.62)
  Figure Delayed Recall pre | 3.28 (4.41) | 14.50 (7.86)
  Figure Delayed Recall post | 7.81 (4.52) | 18.25 (3.25)

6. Primary Outcome: Neurophysiological Function Pre- & Post- Intervention
Description: Resting EEG and ERP recordings before (T1) and after (T2) strengthening exercise intervention
Time Frame: Baseline and 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Early Stage Dementia | Normative Older Adults
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/9
Other Adverse Events (participants affected / at risk) | 0/13 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes